CLINICAL TRIAL: NCT00949546
Title: Treatment of Hidradenitis Suppirativa With Etanercept Injection
Brief Title: Treatment of Hidradenitis Suppurativa Using Etanercept
Status: Completed | Type: Observational
Sponsor: Penn State University (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20031168
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Etanercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- placebo controlled: A randomized, double-blind trial of 3 months duration comparing etanercept 50 mg sc twice weekly to placebo in 20 patients with HS. Patients will be randomized with equal allocation to the two treatment groups.
  Interventions: Drug: etanercept

INTERVENTIONS:
Drug: etanercept — etanercept 50 mg sc twice weekly

SUMMARY:
Therapy with etanercept, a TNF inhibitor will reverse the inflammation, symptoms and quality of life and allow healing of HS.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HS for > 6months defined as tender and/or painful, red nodules and/or plaques (confluent nodules) with or without scarring, foul odor, or draining sinuses clinically with HS
* Localizes to skin folds including any of axillx, breast, abdomen and groin
* active disease
* Negative pregnancy test within 7 days before the first dose of study drug
* Sexually active subjects of childbearing potential must agree to use medically acceptable form of contraception during screening and throughout the study

Exclusion Criteria:

* Concurrent active infection including tuberculosis
* Concurrent therapy or therapy 30 days prior with systemic corticosteroids, systemic immunosuppressants, systemic retinoids or ant-TNF agents
* Severe comorbidities (diabetes mellitus requiring insulin, Q F of any severity, MI, unstable angina eectoris, uncontrolled hypertension, oxygendependent severe pulmonary disease, history of cancer *thin 5_ years except cutaneous basal cell or squamous cell carcinoma or in situ cervical carcinoma, history of TB or TB exposure, chronic hepatitis B or C, SLE, history of multiple sclerosis, transverse myelitis, optic neuritis or epilepsy
* Currently enrolled or enrolled within 90 days prior in any trial for treatment of HS
* Known HIV positive
* Contraindication to etanercept as defined in package insert

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chronic HS
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2005-04; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Physician global assessment of HS of clear or mild at week 12 | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: David R Adams, MD, Pharm D, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Derived] Adams DR, Yankura JA, Fogelberg AC, Anderson BE. Treatment of hidradenitis suppurativa with etanercept injection. Arch Dermatol. 2010 May;146(5):501-4. doi: 10.1001/archdermatol.2010.72. PMID 20479297